CLINICAL TRIAL: NCT01088217
Title: Role of Genetics in Idiopathic Pulmonary Fibrosis (IPF)
Acronym: GWAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Collaborators: University of Colorado, Denver (Other); Vanderbilt University (Other); Landspitali University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2R01HL097163 (NIH)
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Idiopathic Pulmonary Fibrosis; Familial Pulmonary Fibrosis; Idiopathic Interstitial Pneumonia; Familial Interstitial Pneumonia
Keywords: Idiopathic Pulmonary Fibrosis; Familial Pulmonary Fibrosis; Idiopathic Interstitial Pneumonia; Familial Interstitial Pneumonia; Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, lung tissue, DNA, RNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate inherited genetic factors that play a role in the development of familial pulmonary fibrosis and to identify a group of genes that predispose individuals to develop pulmonary fibrosis. Finding the genes that cause pulmonary fibrosis is the first step at developing better methods for early diagnosis and improved treatment for pulmonary fibrosis. The overall hypothesis is that inherited genetic factors predispose individuals to develop pulmonary fibrosis.

DETAILED DESCRIPTION:
Familial Pulmonary Fibrosis (FPF) is a sub-category of the idiopathic interstitial pneumonias (IIPs). IIPs are progressive lung conditions, with limited treatment options and unknown etiology. Though the IIPs have been associated with both genetic risk factors and environmental exposures, the molecular mechanism underlying disease progression remain poorly understood. This investigation seeks to identify a group of genetic loci that play a role in the development of familial interstitial pneumonia (FIP) or FPF, where 2 or more cases of IIP are seen within a family.

ELIGIBILITY:
Inclusion Criteria:

* Two or more family members with a clinical diagnosis of Idiopathic Pulmonary Fibrosis (IPF) or Idiopathic Interstitial Pneumonia (IIP)
* Additional family members may be eligible to participate if two family members are suspected of or diagnosed as having Idiopathic Pulmonary Fibrosis (IPF) or Idiopathic Interstitial Pneumonia (IIP)

Exclusion Criteria:

* Individuals whose pulmonary fibrosis is due to a known cause rather than idiopathic
* Individuals whose pulmonary fibrosis is due to a broader genetic syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families with two or more individuals diagnosed with Idiopathic Pulmonary Fibrosis (IPF) or Idiopathic Interstitial Pneumonia (IIP)
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2008-07; Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Identify a group of genetic loci that play a role in the development of familial interstitial pneumonia and idiopathic interstitial pneumonia. | 10 years
  The purpose of this study is to investigate inherited genetic factors that play a role in the development of pulmonary fibrosis and to identify a group of genetic loci/genes that predispose individuals to develop IIP. We will achieve this goal by employing various methods of genetic technology for gene discovery.

SECONDARY OUTCOMES:
Develop biomarkers using proteomic and genomic approaches that will facilitate establishing the diagnosis and prognosis of both familial and sporadic forms of idiopathic interstitial pneumonia (IIP). | 10 years
  A peripheral blood biomarker or biological signature (gene or protein expression pattern) of idiopathic interstitial pneumonias (IIPs) will simplify and improve the accuracy of diagnosis of IIP and diagnose individuals at an earlier, more treatable, stage of their disease. A peripheral blood biomarker for the diagnosis of IIPs and other interstitial lung diseases (ILDs) will potentially decrease the need for invasive surgical lung biopsy, and thereby avoid the additional cost, morbidity, and mortality associated with surgical lung biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Schwartz, MD, Principal Investigator — University of Colorado Denver; National Jewish Health
Locations (4):
- United States (3):
  - University of Colorado Denver, Aurora, Colorado
  - National Jewish Health and University of Colorado Denver, Denver, Colorado
  - Vanderbilt University, Nashville, Tennessee
- Landspitali University Hospital, Reykjavik, Iceland

REFERENCES:
- See also: Click here to learn more about Familial Pulmonary Fibrosis and this study. — http://medschool.ucdenver.edu/fpf